CLINICAL TRIAL: NCT02665741
Title: Comparison of Colon Adenoma Detection Rate Using Two Distal Colonoscope Attachments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 797109
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Results first posted 2020-06-18 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Colon Cancer Screening; Colon Polyps; Colon Adenomas; Water Exchange Colonoscopy
Keywords: distal colonoscope attachments, colon cancer screening, screening colonoscopy, adenoma detection
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Other): Standard colonoscopy - no distal colonoscope attachment will be used in this arm
  Interventions: Device: Control
- Olympus transparent cap (Experimental): The Olympus transparent cap will be attached to the distal end of colonoscope prior to starting the procedure
  Interventions: Device: Olympus transparent cap
- Medivators Endocuff (Experimental): The Medivators Endocuff will be attached to the distal end of colonoscope prior to starting the procedure
  Interventions: Device: Medivators Endocuff

INTERVENTIONS:
Device: Olympus transparent cap — distal colonoscope attachment
  Arms: Olympus transparent cap
Device: Medivators Endocuff — distal colonoscope attachment
  Arms: Medivators Endocuff
Device: Control — No distal colonoscope attachments
  Arms: Control

SUMMARY:
The goal of this study is to compare two FDA approved distal colonoscope attachment devices, in order to identify which device can increase adenoma detection rate the most without increasing procedure time or risk.

DETAILED DESCRIPTION:
Although mortality from colon cancer is decreasing, it remains the second leading cause of cancer related death in the United States. There are multiple factors contributing to this decrease, such as increased awareness, improving screening techniques, etc.

Of the available modalities approved for colon cancer screening in the United States, colonoscopy is considered the gold standard. Colonoscopy has the advantage of being both diagnostic and therapeutic, allowing the removal of pre-cancerous polyps, before the polyps can transform into cancer. Colonic polyps can occur at any location from the rectum to the cecum. Colonoscopy has been shown to be more effective in decreasing incidence of cancer in the left colon but remains limited in the detection of right sided polyps /lesions 2. This difference based on location is thought to be due to several reasons. Typically the right side of the colon is less clean than the left side during colonoscopy, thereby impairing visualization of polyps. This problem has been overcome by incorporating a "split bowel preparation", which has not become standard of care. However, the problem of not being able to visualize polyps behind folds seen in the colon persists despite improvements in the quality of cleansing of the colon. Various endoscopic technologies have been introduced with the goal of assisting with the manipulation of such colonic folds, and thereby reducing chances of missing polyps behind fold. Two such colonoscope assisted devices including the distal transparent cap and the Endocuff endoscopic overtube.

The Endocuff overtube is a small device with flexible arms arranged in 2 rows. Each row has 8 short, soft arms projecting away from the device. These arms are used to peel back the colonic folds without causing physical damage to enable visualization behind colonic folds. The use of Endocuff overtube has shown promising results in terms of cecal intubation rate and time as well as adenoma detection rates 3.

The transparent cap attachment is a clear plastic device that fits at the end of the colonoscope and extends a short distance past the tip of the colonoscope. It aids in the manipulation of folds and in maintaining a suitable distance from the mucosa, with the goal of improving visualization. Although some studies comparing cap fitted colonoscopy to standard (non- attachment) colonoscopies have shown improved adenoma detection 4, others have shown no significant benefit 5.

Although, these devices have been compared with conventional colonoscopies (i.e without any distal attachment), to the investigator's knowledge, there are currently no studies that have compared these two distal colonoscope attachment devices head-to-head, and none has specifically evaluated effects on detection of right sided adenomas. Also, here at UCDavis, these devices are being used specifically in diagnostic colonoscopies for removal of large polyps and the choice of which specific device is used depends on level of comfort of the advanced endoscopist. The endoscopists participating in the investigators' study do not currently use these devices as part of their routine colonoscopies, thus it is important to provide head to head comparison of these devices to help guide management practice.

Therefore, the investigators' goal is to compare the Endocuff overtube assisted, transparent cap fitted, and non-cap fitted (standard) colonoscopy in patients presenting to UC Davis Medical Center for screening colonoscopies.

In addition, 2 of the 3 investigators will employ the water exchange method during for all arms of the trial, while the other investigator will employ the conventional air method of colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* At least 50 years old
* Presenting for a screening or surveillance colonoscopy at UC Davis Endoscopy Suites

Exclusion Criteria:

* Age less than 50 years
* Prior history of colon cancer
* Patients with inflammatory bowel disease
* Patients suspected to have colon cancer based on non invasive tests such as stool tests for hemoglobin or DNA, or imaging finding suggestive of colon cancer (CT or barium enema).
* Patients undergoing colonoscopy for evaluation of symptoms such as abdominal pain, rectal bleeding, diarrhea, constipation, etc, or patient with iron deficiency anemia suspected to be due to ongoing bleeding inside the colon
* Patients with family history of colon cancer in 1st degree relative below the age of 60
* Patients with family history of hereditary polyposis syndromes such as Lynch syndrome, familial adenomatous polyposis etc, which are associated with an increased risk of colon cancer
* Patients unable to consent
* Pregnant patients
* Incarcerated patients
* Non-English speakers

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Brenner H, Hoffmeister M, Arndt V, Stegmaier C, Altenhofen L, Haug U. Protection from right- and left-sided colorectal neoplasms after colonoscopy: population-based study. J Natl Cancer Inst. 2010 Jan 20;102(2):89-95. doi: 10.1093/jnci/djp436. Epub 2009 Dec 30. PMID 20042716
- [Background] Pioche M, Matsumoto M, Takamaru H, Sakamoto T, Nakajima T, Matsuda T, Abe S, Kakugawa Y, Otake Y, Saito Y. Endocuff-assisted colonoscopy increases polyp detection rate: a simulated randomized study involving an anatomic colorectal model and 32 international endoscopists. Surg Endosc. 2016 Jan;30(1):288-95. doi: 10.1007/s00464-015-4208-8. Epub 2015 Apr 11. PMID 25861907
- [Background] Westwood DA, Alexakis N, Connor SJ. Transparent cap-assisted colonoscopy versus standard adult colonoscopy: a systematic review and meta-analysis. Dis Colon Rectum. 2012 Feb;55(2):218-25. doi: 10.1097/DCR.0b013e31823461ef. PMID 22228167
- [Background] Harada Y, Hirasawa D, Fujita N, Noda Y, Kobayashi G, Ishida K, Yonechi M, Ito K, Suzuki T, Sugawara T, Horaguchi J, Takasawa O, Obana T, Oohira T, Onochi K, Kanno Y, Kuroha M, Iwai W. Impact of a transparent hood on the performance of total colonoscopy: a randomized controlled trial. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):637-44. doi: 10.1016/j.gie.2008.08.029. PMID 19251004

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: No distal colonoscope attachment will be used in this arm
  Control: No distal colonoscope attachments
Period: Overall Study
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
Started | 42 | 42 | 42
Completed | 42 | 42 | 42
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff | Total
Number analyzed (Participants) | 42 | 42 | 42 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.3 (7.4) | 60.0 (6.7) | 60.0 (6.8) | 60 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 18 | 19 | 56
  Male | 23 | 24 | 23 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 3
  White | 31 | 33 | 32 | 96
  More than one race | 5 | 2 | 6 | 13
  Unknown or Not Reported | 2 | 5 | 1 | 8
Smoking status [Count of Participants; unit: Participants]
  Never Smoker | 30 | 24 | 28 | 82
  Former Smoker | 11 | 16 | 13 | 40
  Current Smoker | 1 | 2 | 1 | 4
Alcoholic drinks per week [Mean (Standard Deviation); unit: drinks per week] | 4.0 (3.6) | 6.8 (10.7) | 4.4 (4.0) | 5.07 (6.97)
Diabetes [Count of Participants; unit: Participants] | 4 | 3 | 5 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (4.3) | 28.3 (5.5) | 27.4 (5.4) | 28.07 (5.08)

OUTCOME MEASURES:

1. Primary Outcome: Adenoma Detection Rate
Description: The investigators will compare adenoma detection rate at completion of study across the 3 arms
Time Frame: Completion of procedure
Measure: Number; unit: percentage of adenomas detected
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
Number analyzed (Participants) | 42 | 42 | 42
percentage of adenomas detected | 52.4 | 40.5 | 54.8

2. Secondary Outcome: Proximal Adenoma Detection Rate
Description: The investigators will compare proximal adenoma detection rate at completion of study across the 3 arms
Time Frame: Completion of procedure
Measure: Number; unit: percentage of proximal adenomas
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
Number analyzed (Participants) | 42 | 42 | 42
percentage of proximal adenomas | 45.2 | 35.7 | 50.0

3. Secondary Outcome: Cecal Intubation Rate
Description: The investigators will compare cecal intubation rate at completion of study across the 3 arms
Time Frame: Completion of procedure
Measure: Number; unit: percentage of cecal intubation
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
Number analyzed (Participants) | 42 | 42 | 42
percentage of cecal intubation | 100 | 100 | 100

4. Secondary Outcome: Withdrawal Time
Description: The investigators will compare colonoscopy withdrawal time rate at completion of study across the 3 arms
Time Frame: Completion of procedure
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
Number analyzed (Participants) | 42 | 42 | 42
minutes | 12.9 (5.2) | 12.4 (5.6) | 13.0 (6.2)

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Control | Olympus Transparent Cap | Medivators Endocuff
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/42 | 0/42 | 2/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=42) | Olympus Transparent Cap (N=42) | Medivators Endocuff (N=42)
Bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) — Post polypectomy bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-08): https://cdn.clinicaltrials.gov/large-docs/41/NCT02665741/Prot_SAP_000.pdf